CLINICAL TRIAL: NCT06462430
Title: Genotype-phenotype Correlations of Pediatric Patients With PTEN Hamartoma Tumor Syndrome (PHTS) and Creation of Patient Registry
Brief Title: PTEN Hamartoma Tumor Syndrome Pediatric Patient Registry
Status: Recruiting | Type: Observational
Sponsor: Yale University (Other)
Collaborators: Boston Children's Hospital (Other); Ege University (Other)
Responsible Party: Sponsor
Other Study IDs: 08.11.2022 / 2022-22-02
Record Dates: First submitted 2024-06-12; First posted 2024-06-17 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: PTEN Hamartoma Tumor Syndrome; Macrocephaly Autism Syndrome
Keywords: Phosphotase and tension holomog; Macrocephaly; Autism; PTEN
MeSH Terms: conditions — Hamartoma Syndrome, Multiple; Macrocephaly Autism Syndrome; Megalencephaly; Autistic Disorder

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
PtenTurkiye.org' is a national ( Turkish), web-based registry for PTEN Hamartoma Tumour ( PHTS) syndrome established in 2022. It is designed to increase awareness, gather scientific knowledge by collaboration and increase data accessibility, collect high-quality data on the epidemiology, genetic background and natural history of PHTS especially for pediatric patients so that more accurate follow up guidelines can be recommended.

DETAILED DESCRIPTION:
There is a limited understanding of the natural history of childhood-onset PTEN Hamartoma Tumour Syndrome (PHTS) as a cancer predisposition syndrome. Patient registries are important for longitudinal follow up of these patients. Our aim is to create a Turkish registry especially for pediatric PHTS patients, but registry is open to adult PHTS patients as well.

The purpose is to engage families with children with PHTS in the data-sharing process to accelerate research and drug development and share their experiences with other families as a support if they agree to do so. The registry is open to both adults and children with PHTS.

Most pediatric patients with PHTS have autism spectrum disorders, developmental delays and/or intellectual deficiencies. Patient registry will help us see if they are getting appropriate behaviour interventions. There is no consensus on the guidelines for cancer surveillance in children. The investigators will follow these patients according to 'pediatric follow-up protocol for PTEN (Phosphatase and tensin homolog) mutated children' created by Ciaccio et al. Patient registry will also help if these guidelines are sufficient or need improvements.

Once the individual or their parent/guardian has consented to participate in the registry, the researchers will collect their past and current medical, familial, and other necessary demographic information from their medical records and face to face interviews. The investigators will follow up patients every 6 months or earlier if needed. The investigators will do thorough physical and dysmorphological exam (using autism research exchange dysmorphology check list). For patients with autism and other behavioral problems, the investigators will refer them to child and adolescent psychiatry clinics for evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have clinical findings of PHTS and have mutation in PTEN gene ( VUS included if show clinical findings) and agree to participate in the study

Exclusion Criteria:

* Patients who do not have clinical findings of PHTS and do not have mutation in PTEN gene and do not agree to participate in the study

Min Age: 1 Year | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients living in Türkiye from age 1 to onwards with both genetic and clinical diagnosis of PTEN Hamartoma Tumor syndrome
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Genotype-phenotype correlations of pediatric patients with PTEN Hamartoma Tumor Syndrome (PHTS) and creation of patient registry | 3 years
  Longitudinal follow up of pediatric patients with PTEN Hamartoma Tumor syndrome ( PHTS) and their adult relatives with PHTS for 3 years to better understand this syndrome to be able to find better follow up guidelines.

CONTACTS AND LOCATIONS:
Overall Officials: Hande Kaymakcalan Celebiler, MD, Principal Investigator — Yale University
Locations (1):
- Dr.Canan Kocaman pediatric clinic, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Results of the data
Supporting Information: Study Protocol, CSR
Time Frame: After the results is published
Access Criteria: Researchers need to directly contact the principal investigator to discuss this
URL: https://ptenturkiye.org/